CLINICAL TRIAL: NCT03076944
Title: Evaluation of Desensitization Protocols in Reduction of Dentin Hypersensitivity: A Randomized Clinical Trial
Brief Title: Evaluation of Desensitization Protocols in Reduction of Dentin Hypersensitivity
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Federal University of Uberlandia (Other)
Collaborators: Coordenação de Aperfeiçoamento de Pessoal de Nível Superior. (Other Government); Fundação de Amparo à Pesquisa do estado de Minas Gerais (Other)
Responsible Party: Principal Investigator, PAULO VINICIUS SOARES, Professor, Federal University of Uberlandia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CAAE:60751416.1.0000.5152
Record Dates: First submitted 2017-03-07; First posted 2017-03-10 (Actual); Last update posted 2017-03-29 (Actual); Status verified 2017-03

CONDITIONS: Hypersensitivity Dentin; Dentin Sensitivity; Dentin Hypersensitivity; Dentine Hypersensitivity
MeSH Terms: conditions — Dentin Sensitivity | interventions — UltraEZ

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Neural agent (Active Comparator): UltraEZ. Prophylaxis of the teeth; an application every 48 hours; 4 sessions
  Interventions: Drug: UltraEZ
- Obliterator agent (Active Comparator): Enamelast. Prophylaxis of the teeth; an application every 48 hours; 4 sessions
  Interventions: Drug: Enamelast
- Associative approach (Active Comparator): UltraEZ and Enamelast. Prophylaxis of the teeth; an application every 48 hours; 4 sessions. In each session, fistly the UltraEZ (neural agent) will be applied and after the Enamelast (obliterator agent.)
  Interventions: Drug: UltraEZ; Drug: Enamelast

INTERVENTIONS:
Drug: UltraEZ — Prophylaxis, apply uniformly on the teeth, wait 15 minutes, remove the gel from the teeth with cotton and abundant water.
  Arms: Associative approach; Neural agent
Drug: Enamelast — Prophylaxis; dry the teeth; apply uniformly on the teeth with a thin layer.
  Arms: Associative approach; Obliterator agent

SUMMARY:
The aim of this study is through a double blind randomized clinical trial, evaluate the effectiveness of different clinical protocols in the reduction of dentin hypersensitivity. The desensitization approach (single agent or associated agents) and the long-term effectiveness (baseline, 1 week, 2 weeks, 4 weeks, 12 weeks and 24 weeks) will be evaluated. Data will be collected, tabulated and submitted to statistical analysis.

DETAILED DESCRIPTION:
Dentin hypersensitivity is characterized as an acute and short-term pain with multifactorial etiology. This condition is a clinical challenge due to the different treatment protocols available. Therefore, the aim of this study is through a double blind randomized clinical trial, evaluate the effectiveness of different clinical protocols in the reduction of dentin hypersensitivity. Thirty-two patients with dentin hypersensitivity in at least three teeth will be selected.The teeth will be randomly divided into two different groups according to the desensitization approach (single agent with neural action; single agent with obliterating action; associated technique (neural and obliterator agents). The dentin hypersensitivity level will be evaluated immediately after desensitization and after 1, 2, 4,12 and 24 weeks. Data will be collected, tabulated and submitted to statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

* Healthy individuals
* Both genres, interested in the treatment of Dentin Hypersensitivity
* Patients with all teeth in their mouth
* Patients who have at least three teeth with Dentin hypersensitivity in different quadrants
* Good oral hygiene

Exclusion Criteria:

* Caries or unsatisfactory restorations
* Presence of periodontal disease and or parafunctional habits
* Cracks or enamel fractures
* Extensive or unsatisfactory restorations
* Recent restorations involving the labial surface
* Pulpitis
* Dentures
* Orthodontics
* Smokers
* Pregnant women
* Gastroesophageal disease presence
* Uncontrolled systemic disease
* Severe bruxism
* Constant use of analgesic
* Allergic response to dental products

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Estimated)
Dates: Start 2017-03-20 (Actual); Primary Completion 2017-11 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
Level of cervical dentin hypersensitivity by using visual analog scale | 24 weeks
  Evaluation of the reduction in dentin hypersensitivity levels by using visual analog scale with a 24 weeks follow up.

CONTACTS AND LOCATIONS:
Overall Officials: Paulo V Soares, DDS, MS, PHD, Principal Investigator — Federal University of Uberlandia
Locations (1):
- Federal University of Uberlândia, Uberlândia, Minas Gerais, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Orchardson R, Gangarosa LP Sr, Holland GR, Pashley DH, Trowbridge HO, Ashley FP, Kleinberg I, Zappa U. Dentine hypersensitivity-into the 21st century. Arch Oral Biol. 1994;39 Suppl:113S-119S. doi: 10.1016/0003-9969(94)90197-x. No abstract available. PMID 7702459
- [Background] Davari A, Ataei E, Assarzadeh H. Dentin hypersensitivity: etiology, diagnosis and treatment; a literature review. J Dent (Shiraz). 2013 Sep;14(3):136-45. PMID 24724135
- [Background] Canadian Advisory Board on Dentin Hypersensitivity. Consensus-based recommendations for the diagnosis and management of dentin hypersensitivity. J Can Dent Assoc. 2003 Apr;69(4):221-6. PMID 12662460
- [Background] Brannstrom M. Sensitivity of dentine. Oral Surg Oral Med Oral Pathol. 1966 Apr;21(4):517-26. doi: 10.1016/0030-4220(66)90411-7. No abstract available. PMID 5218158
- [Background] Grippo JO, Simring M, Coleman TA. Abfraction, abrasion, biocorrosion, and the enigma of noncarious cervical lesions: a 20-year perspective. J Esthet Restor Dent. 2012 Feb;24(1):10-23. doi: 10.1111/j.1708-8240.2011.00487.x. Epub 2011 Nov 17. PMID 22296690